CLINICAL TRIAL: NCT07194343
Title: Multicenter Study on Levator Ani Muscle Fixation in Laparoscopic Colposacropexy (FIMEA Multicenter Study)
Brief Title: Posterior Mesh Fixation at the Levator Ani Level in Apical Pelvic Organ Prolapse
Acronym: FIMEA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Collaborators: Carlos III Health Institute (Other Government); Ministry of Science and Innovation, Spain (Other Government)
Responsible Party: Principal Investigator, IRENE MORA HERVAS, Coordinator of the Pelvic Floor Functional Unit at the Hospital de la Santa Creu i Sant Pau, Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PI21/00852
Record Dates: First submitted 2025-09-12; First posted 2025-09-26 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2025-11

CONDITIONS: Prolapse Genital; Prolapse Uterovaginal; Prolapse; Female
Keywords: pelvic organ prolapse; apical prolapse; laparoscopic colposacropexy; mesh fixation; levator ani muscle; surgical outcomes; functional outcomes; anatomical outcomes; sexual function
MeSH Terms: conditions — Prolapse; Pelvic Organ Prolapse

STUDY DESIGN:
Intervention Model Description: Group A: Laparoscopic colposacropexy with posterior mesh fixation to the levator ani muscle (standard technique).
  Group B: Laparoscopic colposacropexy with posterior mesh fixation to the vaginal cuff or cervix, without rectovaginal space dissection (simplified technique).
Who Masked: Participant, Outcomes Assessor
Masking Description: Due to the nature of the surgical intervention, a double-blind design is not feasible. However, the assessment of anatomical and functional outcomes during follow-up will be performed by an evaluator who is blinded to the type of surgical technique used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Standard laparoscopic colposacropexy (Active Comparator): The procedure is based on the laparoscopic colposacropexy technique described by Wattiez in 2001 (Clermont-Ferrand group).
  The standard technique includes dissection of the sacral promontory, the vesicovaginal space, and the rectovaginal space with bilateral pararectal fossae.
  In the vesicovaginal space, the mesh is anchored deeply at the level of the vesical neck, and posteriorly, in the rectovaginal and pararectal spaces, at the level of the levator ani muscle.
  Interventions: Procedure: Laparoscopic colposacropexy with levator ani muscle mesh fixation
- Group B: Simplified laparoscopic colposacropexy (Experimental): The simplified technique includes dissection of the sacral promontory and the vesicovaginal space, but does not involve dissection of the rectovaginal space or the pararectal fossae. In this technique, the posterior mesh is anchored to the posterior aspect of the vaginal vault or cervix. Mesh fixation at the sacral promontory and in the vesicovaginal space is performed within the same anatomical boundaries as in the standard technique.
  Interventions: Procedure: Simplified modification of laparoscopic colposacropexy

INTERVENTIONS:
Procedure: Laparoscopic colposacropexy with levator ani muscle mesh fixation — The standard technique includes dissection of the rectovaginal space and bilateral mesh fixation to the levator ani muscle at the deep limit of the pararectal fossae dissection.
  Arms: Group A: Standard laparoscopic colposacropexy
Procedure: Simplified modification of laparoscopic colposacropexy — Rectovaginal dissection is avoided, and the mesh is anchored to the posterior aspect of the cervix or vaginal vault rather than to the levator ani muscle, representing the specific modification from the standard technique.
  Arms: Group B: Simplified laparoscopic colposacropexy

SUMMARY:
This is a prospective, randomized, multicenter, non-inferiority trial including women with stage II-IV apical pelvic organ prolapse (POP), classified according to the POP-Q system. Participants will be randomized into two groups:

Group A: laparoscopic colposacropexy with posterior mesh fixation to the levator ani muscle.

Group B: laparoscopic colposacropexy with posterior mesh fixation to the vaginal cuff/cervix, without dissection of the rectovaginal space.

The objective of the study is to determine whether a simplified colposacropexy technique is non-inferior to the standard procedure in terms of anatomical and functional outcomes.

The primary outcome is anatomical success, defined as a postoperative POP-Q stage 0-I. Secondary outcomes include functional status and sexual function, evaluated using the PFDI-20 and PISQ-12 questionnaires. Data on prolapse anatomy, related symptoms, and sexual function will be collected at baseline and during follow-up visits at 1, 6, and 12 months after surgery.

This study is supported by a national health research grant from the Instituto de Salud Carlos III (ISCIII), Ministry of Science and Innovation, Spain.

DETAILED DESCRIPTION:
This study is a multicenter, randomized, controlled, evaluator-blinded, non-inferiority clinical trial. The null hypothesis is that colposacropexy with posterior mesh fixation to the vaginal vault (without rectovaginal dissection) is associated with an anatomical and/or functional failure rate that is equal to or more than 15% higher than colposacropexy with posterior mesh fixation to the levator ani muscle (deep rectovaginal dissection). A non-inferiority margin of 15% has been selected because smaller differences are not considered clinically relevant.

With this project, the investigators aim to evaluate the outcomes of a simplified colposacropexy technique that avoids dissection of the rectovaginal space and deep pelvic mesh fixation. Demonstrating non-inferiority would imply rejecting the null hypothesis.

The procedure is indicated for women with stage II-IV uterine or vault prolapse according to the POP-Q classification, with or without associated anterior and/or posterior vaginal wall defects. The decision to perform surgery will be made by the gynecologists, independent of trial participation, to ensure that study enrollment does not influence standard surgical indications. Exclusion criteria include previous abdominal or vaginal mesh prolapse reconstructive surgery or POP-Q stage I or asymptomatic prolapse.

Sample size calculations assume a 91% success rate for the standardized procedure (Lee 2014), a non-inferiority margin of 15%, a 95% confidence interval, and 80% statistical power. A total of 166 patients (83 per group) are required, accounting for a 10% dropout rate.

DESCRIPTION OF THE SURGICAL TECHNIQUE

The vesicovaginal dissection and exposure of the sacral promontory will be performed identically in both groups. A predesigned polypropylene mesh will be used, consisting of:

* an apical end for fixation to the sacral promontory,
* two lateral arms shaped like "butterfly wings" to cover and support the anterior and lateral vaginal walls,
* and two lower arms designed for fixation to the levator ani muscle.

Fixation of the mesh to the vagina, sacral promontory, and (when applicable) the levator ani muscle will be performed using nitinol helical mechanical sutures (Spire'it). At the vesicovaginal space, the mesh will be anchored at the anatomical depth corresponding to the vesical neck level in both groups.

The only difference between groups involves the posterior compartment dissection and mesh fixation:

* Group A (standard technique): the posterior arms of the mesh are anchored bilaterally to the levator ani muscle with mechanical sutures.
* Group B (simplified technique): the posterior arms are removed, and the mesh is anchored only to the vaginal vault or cervix with mechanical sutures, without rectovaginal dissection.

ELIGIBILITY:
Inclusion Criteria:

* Women with primary or recurrent apical prolapse (uterine or vaginal vault) stage II-IV according to the POP-Q classification.
* Women with symptomatic POP with indication of reconstructive POP surgery.
* Agreement to comply with all scheduled visits and assessments through 12 months post-surgery.
* Understand and accept the study procedures and sign the informed consent.

Exclusion Criteria:

* History of abdominal reconstructive surgery for pelvic organ prolapse.
* History of vaginal reconstructive surgery for prolapse using mesh.
* Stage I prolapse according to the POP-Q classification, or asymptomatic prolapse.
* Medical contraindication to general anesthesia.
* Patient preference for vaginal surgical treatment.
* Declines participation in the study.
* Patients with disabilities or unable to understand the terms of the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only female participants are eligible, as the condition under study (apical pelvic organ prolapse) occurs exclusively in women.
Enrollment: 190 (Actual)
Dates: Start 2022-10-06 (Actual); Primary Completion 2025-10-31 (Actual); Study Completion 2025-10-31 (Actual)

PRIMARY OUTCOMES:
Difference in anatomical success rate between simplified (Group B) and standard (Group A) laparoscopic colposacropexy. | 12 months after surgery
  Proportion of participants achieving anatomical success, defined as postoperative POP-Q stage 0-I. The primary analysis will test non-inferiority of the simplified technique (Group B) versus the standard technique (Group A). Non-inferiority will be concluded if the lower bound of the two-sided 95% confidence interval for (Success_B - Success_A) is greater than 15% (non-inferiority margin = 15%). POP-Q assessment will be performed using standardized technique by an evaluator blinded to surgical assignment.

SECONDARY OUTCOMES:
Difference in functional outcomes between simplified (Group B) and standard (Group A) laparoscopic colposacropexy. | 12 months after surgery
  Functional outcomes will be assessed by validated questionnaire: Pelvic Floor Distress Inventory-20 (PFDI-20). Scores will be compared between groups to evaluate whether the simplified technique results in inferior functional outcomes compared with the standard technique in women with stage II-IV apical prolapse.
  PFDI-20 consists of 20 items divided into three subdomains:
  * Pelvic Organ Prolapse Distress Inventory (POPDI-6): Score range: 0 to 24.
  * Colorectal-Anal Distress Inventory (CRADI-8): Score range: 0 to 32.
  * Urinary Distress Inventory (UDI-6): Score range: 0 to 24. Each item is scored from 0 (no distress) to 4 (quite a bit of distress). Subdomain scores are calculated by summing the responses within each section. The total PFDI-20 score is the sum of all three subdomains, with a possible global score ranging from 0 to 80. Higher scores indicate greater symptom severity and higher levels of distress caused by pelvic floor disorders.
Difference in sexual outcomes between simplified (Group B) and standard (Group A) laparoscopic colposacropexy. | 12 months after surgery
  Sexual outcomes will be assessed by validated questionnaire: Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire-12 (PISQ-12). Scores will be compared between groups to evaluate whether the simplified technique results in inferior sexual outcomes compared with the standard technique in women with stage II-IV apical prolapse.
  The PISQ-12 is a validated, condition-specific questionnaire used to assess sexual function in women with pelvic organ prolapse and urinary incontinence. It consists of 12 items covering three domains:
  * Behavioral-Emotional Domain
  * Physical Domain
  * Partner-Related Domain Each item is scored on a scale from 0 to 4 and the total PISQ-12 score ranges from 0 to 48. A higher total score reflects better sexual function and quality of sexual life, while lower scores indicate greater sexual dysfunction related to pelvic floor disorders.

CONTACTS AND LOCATIONS:
Locations (6):
- Spain (6):
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona
  - Hospital Universitari Dexeus, Barcelona, Barcelona
  - Hospital Universitari d'Igualada, Igualada, Barcelona
  - Hospital Universitario Infanta Sofia, San Sebastián de los Reyes, Madrid
  - Hospital General Universitario de Valencia, Valencia, Valencia
  - Hospital Clinico Universitario Virgen de la Arrixaca, Murcia

IPD SHARING:
Plan to Share IPD: No
There are no current plans to share individual participant data (IPD). Data use is restricted to the investigators involved in this project, according to the informed consent provided by participants and ethical committee approval.

REFERENCES:
- [Background] Kuroda K, Hamamoto K, Kawamura K, Masunaga A, Horiguchi A, Ito K. Device Selection Contributes to Operative Time Reduction in Laparoscopic Sacrocolpopexy. Gynecol Minim Invasive Ther. 2025 Mar 15;14(2):157-164. doi: 10.4103/gmit.gmit_155_23. eCollection 2025 Apr-Jun. PMID 40521574
- [Background] Schaub M, Lecointre L, Faller E, Boisrame T, Baldauf JJ, Wattiez A, Akladios CY. Laparoscopic Sacral Colpopexy: The "6-Points" Technique. J Minim Invasive Gynecol. 2017 Nov-Dec;24(7):1081-1082. doi: 10.1016/j.jmig.2017.04.003. Epub 2017 Apr 18. PMID 28435129
- [Background] Bataller E, Ros C, Angles S, Gallego M, Espuna-Pons M, Carmona F. Anatomical outcomes 1 year after pelvic organ prolapse surgery in patients with and without a uterus at a high risk of recurrence: a randomised controlled trial comparing laparoscopic sacrocolpopexy/cervicopexy and anterior vaginal mesh. Int Urogynecol J. 2019 Apr;30(4):545-555. doi: 10.1007/s00192-018-3702-7. Epub 2018 Jul 9. PMID 29987345
- [Background] Habib N, Centini G, Pizzoferrato AC, Bui C, Argay I, Bader G. Laparoscopic promontofixation: Where to stop the anterior dissection? Med Hypotheses. 2019 Mar;124:60-63. doi: 10.1016/j.mehy.2019.02.006. Epub 2019 Feb 2. PMID 30798918
- [Background] Cosma S, Petruzzelli P, Chiado Fiorio Tin M, Parisi S, Olearo E, Fassio F, Zizzo R, Danese S, Benedetto C. Simplified laparoscopic sacropexy avoiding deep vaginal dissection. Int J Gynaecol Obstet. 2018 Nov;143(2):239-245. doi: 10.1002/ijgo.12632. Epub 2018 Aug 24. PMID 30076597
- [Background] Moroni RM, Juliato CRT, Cosson M, Giraudet G, Brito LGO. Does sacrocolpopexy present heterogeneity in its surgical technique? A systematic review. Neurourol Urodyn. 2018 Nov;37(8):2335-2345. doi: 10.1002/nau.23764. Epub 2018 Jul 19. PMID 30024069
- [Background] Gluck O, Blaganje M, Veit-Rubin N, Phillips C, Deprest J, O'reilly B, But I, Moore R, Jeffery S, Haddad JM, Deval B. Laparoscopic sacrocolpopexy: A comprehensive literature review on current practice. Eur J Obstet Gynecol Reprod Biol. 2020 Feb;245:94-101. doi: 10.1016/j.ejogrb.2019.12.029. Epub 2019 Dec 26. PMID 31891897
- [Background] Costantini E, Brubaker L, Cervigni M, Matthews CA, O'Reilly BA, Rizk D, Giannitsas K, Maher CF. Sacrocolpopexy for pelvic organ prolapse: evidence-based review and recommendations. Eur J Obstet Gynecol Reprod Biol. 2016 Oct;205:60-5. doi: 10.1016/j.ejogrb.2016.07.503. Epub 2016 Aug 3. PMID 27566224
- [Background] Maher C, Yeung E, Haya N, Christmann-Schmid C, Mowat A, Chen Z, Baessler K. Surgery for women with apical vaginal prolapse. Cochrane Database Syst Rev. 2023 Jul 26;7(7):CD012376. doi: 10.1002/14651858.CD012376.pub2. PMID 37493538